CLINICAL TRIAL: NCT05246072
Title: Effect of Combined Use of Ivermectin and Colchicine in COVID-19 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAMSU R 179 / 2021
Record Dates: First submitted 2022-02-16; First posted 2022-02-18 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Colchicine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ivermectin + colchicine + standard care (Active Comparator): In addition to the local standard of care for COVID 19 patients, the patient will receive:
  Ivermectin + Colchicine
  Interventions: Drug: Ivermectin + colchicine
- Colchicine + standard care (Active Comparator): In addition to the local standard of care for COVID 19 patients, the patient will receive:
  Colchicine
  Interventions: Drug: Colchicine
- standard care (No Intervention): Patients will receive Standard care

INTERVENTIONS:
Drug: Ivermectin + colchicine — In addition to the local standard of care for COVID 19 patients, the patient will receive Ivermectin + colchicine
  Arms: Ivermectin + colchicine + standard care
Drug: Colchicine — In addition to the local standard of care for COVID 19 patients, the patient will receive colchicine
  Arms: Colchicine + standard care

SUMMARY:
The aim of this study will be to investigate the efficacy of use of combination of Ivermectin and colchicine on severity and outcome Of COVID 19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to performing study procedures.
* Currently hospitalized and requiring medical care for non-sever COVID-19.
* One or more of the following: (positive PCR test or positive antibodies) or (CT Chest consistent with COVID19 infection).

Exclusion Criteria:

* Tocilizumab use.
* Mechanical ventilation
* Requirement of oxygen supplementation >8L/min on admission

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
length of oxygen requirement | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided